CLINICAL TRIAL: NCT00548041
Title: Pilot Study to Evaluate a Rapid HIV Testing Program in the Emergency Department
Brief Title: Rapid HIV Testing Program in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11007
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: HIV Infections
Keywords: HIV; Emergency Department; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rapid HIV Tested (Other): Subjects have HIV testing by oral swab performed.
  Interventions: Other: HIV test by oral swab

INTERVENTIONS:
Other: HIV test by oral swab — Eligible subjects underwent rapid HIV testing by oral swab.

SUMMARY:
The purpose of the study is to evaluate the feasibility of a rapid HIV testing program in the Temple University Hospital(TUH)Emergency Department. We hypothesize that a rapid HIV testing program in the TUH Emergency Department is feasible. Patients presenting to the Adult TUH Emergency Department with certain conditions will be offered rapid HIV testing. Testing will be performed by oral swab using the OraQuick Advance test. Patients will receive post-test counseling.

ELIGIBILITY:
Inclusion Criteria:

One of the following conditions:

* Sexually transmitted disease evaluation or prior history of sexually transmitted disease
* Pregnancy
* Clinical condition that suggests possible immunodeficiency
* History of illicit drug use
* History of chronic viral hepatitis
* Patients with unexplained pneumonia or recurrent pneumonia
* Male patients who have a history of sex with men
* Abdominal pain in a sexually active woman or urethritis in a man
* Trauma.
* Age 18 years old or older.

Exclusion Criteria:

* Age less than 18 years.
* None of the above conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Tedaldi, M.D., Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Undergoing Rapid HIV Testing in the ED: Subjects were seen in the ED and had rapid HIV testing performed.
Period: Overall Study
Arm/Group | Subjects Undergoing Rapid HIV Testing in the ED
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Undergoing Rapid HIV Testing in the ED
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Rapid HIV Testing in Emergency Department
Description: Feasibility was assessed as number of participants who were approached and agreed to participate in rapid HIV testing and then had testing completed.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Subjects Undergoing Rapid HIV Testing in the ED
Number analyzed (Participants) | 100
participants | 100

ADVERSE EVENTS:
Arm/Group | Subjects Undergoing HIV Testing in the ED
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Undergoing HIV Testing in the ED (N=0)
Adverse Events were not collected/addressed (Blood and lymphatic system disorders) | 0 (0) — Adverse Events were not collected/assessed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No